CLINICAL TRIAL: NCT00488631
Title: A Phase 3 Multicenter, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Safety and Efficacy of Golimumab Maintenance Therapy, Administered Subcutaneously, in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: An Efficacy and Safety Study of Golimumab (CNTO 148) in Participants With Moderately to Severely Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR014179; 2006-003399-37 (EudraCT Number); C0524T18 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-03

CONDITIONS: Colitis, Ulcerative
Keywords: Colitis, Ulcerative; Golimumab; CNTO 148
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Golimumab induction responders (GLM-I-Rsp)-Placebo Maintenance (Placebo Comparator): Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to placebo subcutaneous (under the skin) injection matching to golimumab administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631). Participants with loss of clinical response will have their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52.
  Interventions: Biological: Placebo; Biological: Golimumab 100 mg
- GLM-I-Rsp-Golimumab 50 mg Maintenance (Experimental): Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to golimumab 50 mg subcutaneous injection administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631). Participants with loss of clinical response will be re-randomized to receive golimumab 50 mg or 100 mg subcutaneous injections every 4 weeks through Week 52.
  Interventions: Biological: Golimumab 50 mg; Biological: Golimumab 100 mg
- GLM-I-Rsp-Golimumab 100 mg Maintenance (Experimental): Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631). Participants with loss of clinical response will be re-randomized to receive golimumab 100 mg or 200 mg subcutaneous injections every 4 weeks through Week 52.
  Interventions: Biological: Golimumab 100 mg; Biological: Golimumab 200 mg
- Placebo induction responders (PBO-I-Rsp)-Placebo Maintenance (Placebo Comparator): Participants in clinical response to placebo at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and received placebo subcutaneous injection matching to golimumab administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631); not randomized. Participants with loss of clinical response will have their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52.
  Interventions: Biological: Placebo; Biological: Golimumab 100 mg
- PBO-I-nonRsp-Golimumab 100 mg Maintenance (Experimental): Participants not in clinical response to placebo at Week 6 induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and received golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631); not randomized.
  Interventions: Biological: Golimumab 100 mg
- GLM-I-nonRsp-Golimumab 100 mg Maintenance (Experimental): Participants not in clinical response to golimumab at Week 6 of induction study and received golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631); not randomized.
  Interventions: Biological: Golimumab 100 mg

INTERVENTIONS:
Biological: Placebo — Participants receive placebo subcutaneous injection matching to golimumab administered every 4 weeks through Week 52 in the maintenance study C0524T18 (NCT00488631).
  Arms: Golimumab induction responders (GLM-I-Rsp)-Placebo Maintenance; Placebo induction responders (PBO-I-Rsp)-Placebo Maintenance
Biological: Golimumab 50 mg — Participants receive golimumab 50 mg subcutaneous injection administered every 4 weeks through Week 52 in the maintenance study C0524T18 (NCT00488631).
  Arms: GLM-I-Rsp-Golimumab 50 mg Maintenance
Biological: Golimumab 100 mg — Participants receive golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52 in the maintenance study C0524T18 (NCT00488631) initially or after dose adjustment following loss of clinical response.
Biological: Golimumab 200 mg — Participants receiving golimumab 100 mg initially who on loss of clinical response receive golimumab 200 mg administered every 4 weeks through Week 52.
  Arms: GLM-I-Rsp-Golimumab 100 mg Maintenance

SUMMARY:
The purpose of this study is to assess the safety and efficacy of golimumab administered subcutaneously (under the skin) injections in maintenance therapy.

DETAILED DESCRIPTION:
This was a Phase 3, multicenter (conducted in more than one center), placebo-controlled (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), double-blind (neither the Physician nor the participant know about the study medication), parallel-group (a medical research study comparing the response in 2 or more groups of participants receiving different interventions), randomized-withdrawal study. Participants who were in clinical response to golimumab at Week 6 in induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) will be randomly assigned in a 1:1:1 ratio at Week 0 of this study to receive 1 of the following maintenance treatment regimens administered subcutaneously every 4 weeks through Week 52: placebo, golimumab 50 mg, or golimumab 100 mg. Participants who were in clinical response to placebo and participants who were not in clinical response to golimumab or placebo at Week 6 in induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) will not be randomly assigned but will be eligible to be enrolled in the study (i.e., the nonrandomized group) and received the following treatment regimens: placebo, golimumab 100 mg and golimumab 100 mg. Dose adjustment will be done for participants who were in clinical response to golimumab or placebo during induction studies C0524T16 (NCT00488774) or C0524T17 (NCT00487539) but lose clinical response during maintenance study C0524T18 (NCT00488631). On completing this study, participant will have the opportunity to continue to receive study medication in a study extension that will last up to approximately 3 years. Efficacy will be primarily evaluated by assessing the clinical response using Mayo Score. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who received all study agent administrations and completed the Week 6 Mayo score evaluation in induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539)
* Participants who completed the Week 0 visit for this maintenance study C0524T18 (NCT00488631) on the same day as the Week 6 visit of the induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539)

Exclusion Criteria:

* Participants who increased the dose of their concomitant (given at the same time) UC medications since Week 0 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539)
* Participants who initiated a concomitant UC medication since Week 0 of an induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539)
* Participants who had a partial or total colectomy (surgery to remove part or all of the colon) or an ostomy (surgical construction of an artificial opening (stoma) for external fistulization of a duct or vessel by insertion of a tube with or without a supportive stent) since Week 0 of an induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539)
* Participants with signs or symptoms of latent or active granulomatous infection (including TB); a nontuberculous mycobacterial infection or opportunistic infection; or infection with HIV (Human Immunodeficiency Virus), hepatitis B, or hepatitis C
* Participants with signs and symptoms of any malignancy or suggestive of a possible lymphoproliferative disease (disorders characterized by proliferation of lymphoid tissue, general or unspecified)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1228 (Actual)
Dates: Start 2007-09; Primary Completion 2011-10 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (297):
- United States (96):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Anaheim, California
  - Merced, California
  - Orange, California
  - Roseville, California
  - San Diego, California
  - Lakewood, Colorado
  - Littleton, Colorado
  - Bristol, Connecticut
  - Newark, Delaware
  - Boca Raton, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - North Miami Beach, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Savannah, Georgia
  - Snellville, Georgia
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Clive, Iowa
  - Fort Dodge, Iowa
  - Pratt, Kansas
  - Topeka, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Monroe, Louisiana
  - Hagerstown, Maryland
  - Hollywood, Maryland
  - Laurel, Maryland
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Dearborn, Michigan
  - Troy, Michigan
  - Plymouth, Minnesota
  - Rochester, Minnesota
  - Pascagoula, Mississippi
  - Tupelo, Mississippi
  - Urbana, Missouri
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Egg Harbor, New Jersey
  - Great Neck, New York
  - Huntington, New York
  - New York, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Boone, North Carolina
  - Charlotte, North Carolina
  - Harrisburg, North Carolina
  - Kinston, North Carolina
  - Morganton, North Carolina
  - New Bern, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Colombus, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Limerick, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Galveston, Texas
  - Houston, Texas
  - Logan, Utah
  - Ogden, Utah
  - Burlington, Vermont
  - Chesapeake, Virginia
  - Christiansburg, Virginia
  - Fairfax, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (13):
  - Adelaide
  - Bankstown
  - Box Hill
  - Brisbane
  - Cairns
  - Fitzroy
  - Fremantle
  - Herston
  - Launceston
  - Malvern
  - Parkville
  - Prahran
  - Westmead
- Austria (2):
  - Innsbruck
  - Vienna
- Belgium (6):
  - Bonheiden
  - Brussels
  - Ghent
  - Leuven
  - Liège
  - Roeselare
- Bulgaria (5):
  - Bulgaria
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
- Canada (15):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Barrie, Ontario
  - Chatham, Ontario
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Vaughan, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan
  - Toronto
  - Windsor
- Czechia (4):
  - Èeské Budìjovice 1
  - Hradec Králové
  - Litoměřice
  - Ostrava
- Denmark (4):
  - Aalborg
  - Aarhus C
  - Hvidovre
  - Odense C
- France (8):
  - Amiens Cedex 1 80
  - Bordeaux
  - Clichy
  - Lille
  - Marseille
  - Nice
  - Paris
  - Rouen
- Germany (17):
  - Aachen
  - Berlin
  - Berlin Be
  - Bochum
  - Frankfurt
  - Hamburg
  - Hanover
  - Heidelberg
  - Herne
  - Jena
  - Kiel
  - Magdeburg
  - Minden
  - München
  - Münster
  - Neustadt
  - Stade
- Hungary (18):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Dunaújváros
  - Gyõr
  - Gyula
  - Gyulai Ut 18
  - Miskolc
  - Mosonmagyaróvár
  - Pécs
  - Siófok
  - Sopron
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Szombathely
  - Veszprém
  - Zalaegerszeg
- India (11):
  - Bangalore
  - Chennai
  - Hyderabad
  - Hyderabad Andh Prad
  - Jaipur
  - Kārnād
  - Lucknow Gpo
  - Ludhiana
  - New Delhi
  - Pune
  - Vishakapatanam
- Israel (13):
  - Afula
  - Beer Yaakov
  - Beersheba
  - Haifa
  - Hedera
  - Jerusalem
  - Kfar Saba
  - Kiryat Bialik
  - Nazareth
  - Petah-Tikv
  - Rehovot
  - Tel Aviv
  - Tel Litwinsky
- Japan (15):
  - Bunkyō City
  - Chikushinoshi
  - Fukuoka
  - Hiroshima
  - Kagoshima
  - Kurashiki
  - Kurume
  - Nagoya
  - Nishinomiya
  - Okayama
  - Osaka
  - Sakura
  - Sapporo
  - Tokyo
  - Yokkaichi
- Latvia (3):
  - Balvi
  - Daugavpils
  - Riga
- Lithuania (5):
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
  - Vilnius Lt
- Netherlands (6):
  - Amsterdam
  - Ede Gld
  - Groningen
  - Leiden
  - Nieuwegein
  - Rotterdam
- New Zealand (5):
  - Auckland
  - Christchurch
  - Dunedin
  - Hamilton
  - Hastings
- Poland (14):
  - Bialystok
  - Bydgoszcz
  - Częstochowa
  - Elblag
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Opole
  - Skierniewice
  - Sopot
  - Szczecin
  - Torun
  - Warsaw
- Romania (5):
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Târgu Mureş
  - Timișoara
- Russia (6):
  - Moscow
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Smolensk
  - Yaroslavl
- Serbia (3):
  - Belgrade
  - Niš
  - Zemun
- Slovakia (6):
  - Bratislava
  - Martin
  - Nitra
  - Nové Mesto nad Váhom
  - Prešov
  - Trnava
- South Africa (5):
  - Cape Town
  - Cape Town West Cape
  - Durban
  - Plumstead West Cape
  - Pretoria Gauteng
- Sweden (2):
  - Gothenburg
  - Stockholm
- Ukraine (10):
  - Donetsk
  - Ivano
  - Kharkiv
  - Kiev
  - Kyiv
  - Lviv
  - Poltava
  - Simferopol
  - Vinnitsa
  - Zhaporozhia 69104

REFERENCES:
- [Derived] Weinstein CLJ, Meehan AG, Govoni M, Lin J, Reinisch W. Low Occurrence of Colectomy With Long-Term (up to 4 Years) Golimumab Treatment in Patients With Moderate-to-Severe Active Ulcerative Colitis: Data From the PURSUIT Maintenance and Long-Term Extension Studies. Crohns Colitis 360. 2023 Aug 26;5(3):otad044. doi: 10.1093/crocol/otad044. eCollection 2023 Jul. PMID 37691729
- [Derived] Perrig K, Krupka N, Jordi SBU, Rossel JB, Biedermann L, Greuter T, Schreiner P, Vavricka SR, Juillerat P, Burri E, Zimmermann D, Maillard MH, Sulz MC, Brand S, Rogler G, Misselwitz B. Effectiveness of golimumab in patients with ulcerative colitis: results of a real-life study in Switzerland. Therap Adv Gastroenterol. 2022 Feb 9;15:17562848221074188. doi: 10.1177/17562848221074188. eCollection 2022. PMID 35154389
- [Derived] Adedokun OJ, Xu Z, Liao S, Strauss R, Reinisch W, Feagan BG, Sandborn WJ. Population Pharmacokinetics and Exposure-Response Modeling of Golimumab in Adults With Moderately to Severely Active Ulcerative Colitis. Clin Ther. 2020 Jan;42(1):157-174.e4. doi: 10.1016/j.clinthera.2019.11.010. Epub 2020 Jan 22. PMID 31982148
- [Derived] Philip G, Cornillie F, Adedokun JO, Melsheimer R, Rutgeerts P, Colombel JF, Marano C. Early Dose Optimisation of Golimumab in Nonresponders to Induction Treatment for Ulcerative Colitis Is Effective and Supported by Pharmacokinetic Data. J Crohns Colitis. 2019 Sep 27;13(10):1257-1264. doi: 10.1093/ecco-jcc/jjz052. PMID 30847474
- [Derived] Reinisch W, Gibson PR, Sandborn WJ, Feagan BG, Strauss R, Johanns J, Padgett L, Adedokun OJ, Colombel JF, Collins J, Rutgeerts P, Tarabar D, Marano C. Long-Term Benefit of Golimumab for Patients with Moderately to Severely Active Ulcerative Colitis: Results from the PURSUIT-Maintenance Extension. J Crohns Colitis. 2018 Aug 29;12(9):1053-1066. doi: 10.1093/ecco-jcc/jjy079. PMID 29917070
- [Derived] Sandborn WJ, Feagan BG, Marano C, Zhang H, Strauss R, Johanns J, Adedokun OJ, Guzzo C, Colombel JF, Reinisch W, Gibson PR, Collins J, Jarnerot G, Rutgeerts P; PURSUIT-Maintenance Study Group. Subcutaneous golimumab maintains clinical response in patients with moderate-to-severe ulcerative colitis. Gastroenterology. 2014 Jan;146(1):96-109.e1. doi: 10.1053/j.gastro.2013.06.010. Epub 2013 Jun 14. PMID 23770005

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Efficacy results are based on participants who were Golimumab induction responders (GLM-I-Rsp) and were randomly assigned to GLM-I-Rsp-Placebo Maintenance, GLM-I-Rsp-Golimumab 50 mg and GLM-I-Rsp-Golimumab 100 mg as per planned analysis.
Groups:
- Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance: Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to placebo subcutaneous injection matching to golimumab administered every 4 weeks through Week 52 in the maintenance study C0524T18 (NCT00488631). Participants with loss of clinical response had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52. For participants with dose adjustment, adverse events are presented from Week 0 up to the time of dose adjustment.
- GLM-I-Rsp-Golimumab 50 mg Maintenance: Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to golimumab 50 mg subcutaneous injection administered every 4 weeks through Week 52 in C0524T18 (NCT00488631). Participants with loss of clinical response were re-randomized to receive golimumab 50 mg or 100 mg subcutaneous injection administered every 4 weeks through Week 52. For participants with dose adjustment, adverse events are presented from Week 0 up to the time of dose increase.
- GLM-I-Rsp-Golimumab 100 mg Maintenance: Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631). Participants with loss of clinical response were re-randomized to receive golimumab 100 mg or 200 mg subcutaneous injection administered every 4 weeks through Week 52 (prior to protocol amendment 3). For participants with dose adjustment, adverse events are presented from Week 0 up to the time of dose increase.
- Placebo Induction Responders (PBO-I-Rsp)-Placebo Maintenance: Participants in clinical response to placebo at Week 6 of an induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and received placebo subcutaneous injection matching to golimumab every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631); not randomized. Participants with loss of clinical response had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52. For participants with dose adjustment, adverse events are presented from Week 0 up to the time of dose adjustment.
- PBO-I-nonRsp-Golimumab 100 mg Maintenance: Participants not in clinical response to placebo at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and received golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631); not randomized.
- GLM-I-nonRsp-Golimumab 100 mg Maintenance: Participants not in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and received golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631); not randomized.
- Placebo Extension: Participants entered the study extension at Week 54 receiving placebo subcutaneous injection administered every 4 weeks until study unblinding and discontinuation of participants remaining on placebo; those whose UC disease worsened had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks in the study extension.
- Golimumab 50 mg - Extension: Participants entered the study extension at Week 54 receiving golimumab 50 mg subcutaneous injection administered every 4 weeks; those whose UC disease worsened had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks.
- Golimumab 100 mg Extension: Participants entered the study extension at Week 54 receiving golimumab 100 mg subcutaneous injection administered every 4 weeks; prior to Amendment 3 , those whose UC disease worsened had their dose increased to golimumab 200 mg subcutaneous injection administered every 4 weeks.
- Golimumab 200 mg Extension: Participants entered the study extension at Week 54 receiving golimumab 200 mg subcutaneous injection administered every 4 weeks. With Amendment 3 participants remaining on golimumab 200 mg had their dose decreased to golimumab 100 mg subcutaneous injection administered every 4 weeks.
Period: Double Blind Period (Week 0-54)
Arm/Group | Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance | GLM-I-Rsp-Golimumab 50 mg Maintenance | GLM-I-Rsp-Golimumab 100 mg Maintenance | Placebo Induction Responders (PBO-I-Rsp)-Placebo Maintenance | PBO-I-nonRsp-Golimumab 100 mg Maintenance | GLM-I-nonRsp-Golimumab 100 mg Maintenance | Placebo Extension | Golimumab 50 mg - Extension | Golimumab 100 mg Extension | Golimumab 200 mg Extension
Started | 156 | 154 | 154 | 129 | 230 | 405 | 0 | 0 | 0 | 0
Completed | 113 | 111 | 109 | 88 | 127 | 189 | 0 | 0 | 0 | 0
Not Completed | 43 | 43 | 45 | 41 | 103 | 216 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 17 | 12 | 12 | 12 | 30 | 50 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 19 | 17 | 22 | 18 | 56 | 124 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 3 | 7 | 0 | 0 | 0 | 0
Not completed — Other | 6 | 12 | 10 | 11 | 14 | 34 | 0 | 0 | 0 | 0
Period: Open Label Study Extension (Week 54-228)
Arm/Group | Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance | GLM-I-Rsp-Golimumab 50 mg Maintenance | GLM-I-Rsp-Golimumab 100 mg Maintenance | Placebo Induction Responders (PBO-I-Rsp)-Placebo Maintenance | PBO-I-nonRsp-Golimumab 100 mg Maintenance | GLM-I-nonRsp-Golimumab 100 mg Maintenance | Placebo Extension | Golimumab 50 mg - Extension | Golimumab 100 mg Extension | Golimumab 200 mg Extension
Started | 0 | 0 | 0 | 0 | 0 | 0 | 96 | 93 | 470 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 66 | 288 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 80 | 27 | 182 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 8 | 54 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 34 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 0
Not completed — Unspecified reasons | 0 | 0 | 0 | 0 | 0 | 0 | 63 | 14 | 87 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance | GLM-I-Rsp-Golimumab 50 mg Maintenance | GLM-I-Rsp-Golimumab 100 mg Maintenance | Placebo Induction Responders (PBO-I-Rsp)-Placebo Maintenance | PBO-I-nonRsp-Golimumab 100 mg Maintenance | GLM-I-nonRsp-Golimumab 100 mg Maintenance | Total
Number analyzed (Participants) | 156 | 154 | 154 | 129 | 230 | 405 | 1228
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (14.05) | 41.4 (13.84) | 39.1 (13.11) | 38 (13.27) | 40.3 (12.67) | 41.2 (13.6) | 40.3 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 77 | 65 | 68 | 99 | 138 | 528
  Male | 75 | 77 | 89 | 61 | 131 | 267 | 700

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Clinical Response Through Week 54
Description: Clinical response is defined as decrease from induction baseline in Mayo score by greater than or equal to (>=) 30 percent and >= 3, with either decrease from induction baseline in rectal bleeding subscore of >= 1 or rectal bleeding subscore of 0 or 1. Participants who lost clinical response prior to Week 54 were considered not to meet endpoint. Mayo score is sum of 4 subscores (ie, stool frequency, rectal bleeding, endoscopic findings, physician's global assessment); each rated on scale from 0 to 3, with higher scores indicating more severe disease. Total Mayo score value ranges from 0 to 12.
Time Frame: Induction Baseline, Week 0 through Week 54
Population: Primary analysis population included randomly assigned participants in clinical response to golimumab induction at Week 0 of the maintenance study. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Participants
Groups:
- Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance: Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to placebo subcutaneous (under the skin) injection matching to golimumab administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631). Participants with loss of clinical response had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52.
- GLM-I-Rsp-Golimumab 100 mg Maintenance: Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631). Adverse events are presented through Week 54. Participants with loss of clinical response were re-randomized to receive golimumab 100 mg or 200 mg subcutaneous injection administered every 4 weeks through Week 52 (prior to protocol amendment 3). For participants with dose adjustment, adverse events are presented from Week 0 up to the time of dose increase.
Arm/Group | Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance | GLM-I-Rsp-Golimumab 50 mg Maintenance | GLM-I-Rsp-Golimumab 100 mg Maintenance
Number analyzed (Participants) | 154 | 151 | 151
Participants | 48 | 71 | 75
Statistical Analysis 1: Comparison: Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance vs GLM-I-Rsp-Golimumab 50 mg Maintenance; Statistical analysis for number of participants in clinical response through Week 54 were summarized using the Cochran-Mantel-Haenszel (CMH) test stratified by clinical remission status at Week 0 and the induction dose factor; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel — A fixed sequence testing procedure was employed to control the overall Type I error rate at the 0.05 level (i.e., testing golimumab 100 mg vs. placebo first, then, if positive, testing 50 mg vs. placebo)
Statistical Analysis 2: Comparison: Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance vs GLM-I-Rsp-Golimumab 100 mg Maintenance; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Clinical Remission at Both Week 30 and Week 54
Description: Clinical remission is defined as a Mayo score of less than or equal to 2, with no individual sub-score greater than 1. The Mayo score is sum of 4 sub-scores (i.e., stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total Mayo score value ranges from 0 to 12. The number of participants in clinical remission at both the weeks that is Week 30 as well as Week 54 will be reported.
Time Frame: Week 30 and Week 54
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance | GLM-I-Rsp-Golimumab 50 mg Maintenance | GLM-I-Rsp-Golimumab 100 mg Maintenance
Number analyzed (Participants) | 154 | 151 | 151
Participants | 24 | 35 | 42
Statistical Analysis 1: Comparison: Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance vs GLM-I-Rsp-Golimumab 50 mg Maintenance; Statistical analysis for number of participants with clinical remission at both Week 30 and Week 54 were summarized using the CMH test stratified by clinical remission status at Week 0 and the induction dose factor; Test type: Superiority or Other; p = 0.122, Cochran-Mantel-Haenszel — Fixed sequence testing; 100 mg group was tested if it was positive for preceding endpoint, regardless whether 50 mg group was positive;50 mg group was tested if 100 mg group positive for same endpoint and 50 mg group positive for preceding endpoint
Statistical Analysis 2: Comparison: Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance vs GLM-I-Rsp-Golimumab 100 mg Maintenance; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Participants With Mucosal Healing at Both Week 30 and Week 54
Description: Mucosal healing is determined from the endoscopy sub-score of the Mayo score. Mucosal healing is defined as an endoscopy sub-score of 0 or 1. Higher score indicates higher severity of disease. Endoscopy sub-score ranges from 0 (normal or inactive disease) to 3 (severe disease; spontaneous bleeding and ulceration). The number of participants with mucosal healing at both the weeks that is Week 30 as well as Week 54 will be reported.
Time Frame: Week 30 and Week 54
Population: Primary analysis population included randomly assigned participants in clinical response to golimumab induction at Week 0 of the study. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Participants
Arm/Group | Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance | GLM-I-Rsp-Golimumab 50 mg Maintenance | GLM-I-Rsp-Golimumab 100 mg Maintenance
Number analyzed (Participants) | 154 | 151 | 151
Participants | 41 | 63 | 64
Statistical Analysis 1: Comparison: Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance vs GLM-I-Rsp-Golimumab 50 mg Maintenance; Statistical analysis for number of participants with mucosal healing at both Week 30 and Week 54 were summarized using CMH test stratified by clinical remission status at Week 0 and the induction dose factor; Test type: Superiority or Other; p = 0.011, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance vs GLM-I-Rsp-Golimumab 100 mg Maintenance; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Participants With Clinical Remission at Both Week 30 and 54 Among Participants With Clinical Remission at Week 0 of Maintenance Study
Description: as for outcome 2
Time Frame: Week 30 and Week 54
Population: Analysis population included randomly assigned participants who were in clinical remission to golimumab induction at Week 0 of the maintenance study. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Participants
Arm/Group | Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance | GLM-I-Rsp-Golimumab 50 mg Maintenance | GLM-I-Rsp-Golimumab 100 mg Maintenance
Number analyzed (Participants) | 54 | 52 | 54
Participants | 13 | 19 | 21
Statistical Analysis 1: Comparison: Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance vs GLM-I-Rsp-Golimumab 50 mg Maintenance; Statistical analysis for number of participants with clinical remission at both Week 30 and 54 among participants with clinical remission at Week 0 of maintenance study were summarized using CMH test stratified by the induction dose factor; Test type: Superiority or Other; p = 0.365, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance vs GLM-I-Rsp-Golimumab 100 mg Maintenance; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.098, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

5. Secondary Outcome: Number of Participants With Clinical Remission at Week 54 and Not Receiving Concomitant Corticosteroids Among Participants on Corticosteroids at Week 0 of Maintenance Study
Description: Clinical remission is defined as a Mayo score of less than or equal to 2, with no individual sub-score greater than 1. The Mayo score is sum of 4 sub-scores (i.e., stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total Mayo score value ranges from 0 to 12.
Time Frame: Week 54
Population: Analysis population included randomly assigned participants in clinical response to golimumab induction who were receiving concomitant corticosteroids at Week 0 of the study. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Participants
Arm/Group | Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance | GLM-I-Rsp-Golimumab 50 mg Maintenance | GLM-I-Rsp-Golimumab 100 mg Maintenance
Number analyzed (Participants) | 87 | 78 | 82
Participants | 16 | 22 | 19
Statistical Analysis 1: Comparison: Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance vs GLM-I-Rsp-Golimumab 50 mg Maintenance; Statistical analysis for number of participants with clinical remission at Week 54 and not receiving concomitant corticosteroids among participants on corticosteroids at Week 0 of maintenance study were summarized using the CMH test stratified by clinical remission status at Week 0 and the induction dose factor; Test type: Superiority or Other; p = 0.279, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance vs GLM-I-Rsp-Golimumab 100 mg Maintenance; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.423, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Groups:
- Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance: Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to placebo subcutaneous injection matching to golimumab administered every 4 weeks through Week 52 in the maintenance study C0524T18 (NCT00488631). Adverse events are presented through Week 54. Participants with loss of clinical response had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52. For participants with dose adjustment, adverse events are presented from Week 0 up to the time of dose adjustment.
- GLM-I-Rsp-Golimumab 50 mg Maintenance: Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to golimumab 50 mg subcutaneous injection administered every 4 weeks through Week 52 in C0524T18 (NCT00488631). Adverse events are presented through Week 54.Participants with loss of clinical response were re-randomized to receive golimumab 50 mg or 100 mg subcutaneous injection administered every 4 weeks through Week 52. For participants with dose adjustment, adverse events are presented from Week 0 up to the time of dose increase.
- GLM-I-Rsp-Placebo Maintenance-Golimumab 100 mg; GLM-I-Rsp-Golimumab 50 mg Maintenance-Golimumab 100 mg: Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to placebo every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631), and had their dose increased to golimumab 100 mg subcutaneous injection every 4 weeks through Week 52 on loss of clinical response Adverse events are presented from the time of dose adjustment onwards up to Week 54.
- GLM-I-Rsp-Golimumab 100 mg Maintenance-Golimumab 200 mg: Participants in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and randomized to golimumab 100 mg subcutaneous injection every 4 weeks through Week 52 in the maintenance study C0524T18 (NCT00488631), and had their dose increased to golimumab 200 mg subcutaneous injection every 4 weeks through Week 52 on loss of clinical response. Adverse events are presented from the time of dose adjustment onwards up to Week 54.
- Placebo Induction Responders (PBO-I-Rsp)-Placebo Maintenance: Participants in clinical response to placebo at Week 6 of an induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and received placebo subcutaneous injection matching to golimumab every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631); not randomized. Adverse events are presented through Week 54. Participants with loss of clinical response had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52. For participants with dose adjustment, adverse events are presented from Week 0 up to the time of dose adjustment.
- PBO-I-nonRsp-Golimumab 100 mg Maintenance: Participants not in clinical response to placebo at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and received golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631); not randomized. Adverse events are presented through Week 54.
- GLM-I-nonRsp-Golimumab 100 mg Maintenance: Participants not in clinical response to golimumab at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and received golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631); not randomized. Adverse events are presented through Week 54.
- PBO-I-Rsp-Placebo Maintenance-Golimumab 100 mg: Participants in clinical response to placebo at Week 6 of induction study C0524T16 (NCT00488774) or C0524T17 (NCT00487539) and received placebo every 4 weeks through Week 52 in maintenance study C0524T18 (NCT00488631) and had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks through Week 52 on loss of clinical response; not randomized. Adverse events are presented from the time of dose adjustment onwards up to Week 54.
- Placebo Extension: Participants entered the study extension receiving placebo subcutaneous injection administered every 4 weeks until study unblinding and discontinuation of participants remaining on placebo; those whose UC disease worsened had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks in the study extension. Adverse events are presented from Week 54 up to Week 228 or the time of dose adjustment for subjects who increased dose.
- Golimumab 50 mg Extension Phase: Participants entered the study extension receiving golimumab 50 mg subcutaneous injection administered every 4 weeks; those whose UC disease worsened had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks. Adverse events are presented from Week 54 up to Week 228 or the time of dose adjustment for subjects who increased dose.
- Golimumab 100 mg Extension: Participants entered the study extension receiving golimumab 100 mg subcutaneous injection administered every 4 weeks; prior to Amendment 3 , those whose UC disease worsened had their dose increased to golimumab 200 mg subcutaneous injection administered every 4 weeks. Adverse events are presented from Week 54 up to Week 228 or the time of dose adjustment for subjects who increased dose.
- Golimumab 200 mg Extension: Participants entered the study extension receiving golimumab 200 mg subcutaneous injection administered every 4 weeks. With Amendment 3 participants remaining golimumab 200 mg had their dose descreased to golimumab 100 mg subcutaneous injection administered every 4 weeks. Adverse events are presented from Week 54.
- Placebo - 50 mg Extension: A single participant entered the study extension receiving placebo subcutaneous injection administered every 4 weeks; and on worsening of UC disease had their dose increased to golimumab 50 mg subcutaneous injection administered every 4 weeks in the study extension. Adverse events are presented from the time of dose adjustment.
- Placebo - Golimumab100 mg Extension: Participants entered the study extension receiving placebo subcutaneous injection administered every 4 weeks and had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks upon worsening of UC disease in the study extension. Adverse events are presented from the time of dose adjustment.
- Golimumab 50 mg - 100 mg Extension: Participants entered the study extension receiving golimumab 50 mg subcutaneous injection administered every 4 weeks and had their dose increased to golimumab 100 mg subcutaneous injection administered every 4 weeks upon worsening of UC disease. Adverse events are presented from the time of dose adjustment
- Golimumab 100 mg - 200 mg Extension: Participants entered the study extension receiving golimumab 100 mg subcutaneous injection administered every 4 weeks and had their dose increased to golimumab 200 mg subcutaneous injection administered every 4 weeks upon worsening of UC disease. Adverse events are presented from the time of dose adjustment.
Arm/Group | Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance | GLM-I-Rsp-Golimumab 50 mg Maintenance | GLM-I-Rsp-Golimumab 100 mg Maintenance | GLM-I-Rsp-Placebo Maintenance-Golimumab 100 mg | GLM-I-Rsp-Golimumab 50 mg Maintenance-Golimumab 100 mg | GLM-I-Rsp-Golimumab 100 mg Maintenance-Golimumab 200 mg | Placebo Induction Responders (PBO-I-Rsp)-Placebo Maintenance | PBO-I-nonRsp-Golimumab 100 mg Maintenance | GLM-I-nonRsp-Golimumab 100 mg Maintenance | PBO-I-Rsp-Placebo Maintenance-Golimumab 100 mg | Placebo Extension | Golimumab 50 mg Extension Phase | Golimumab 100 mg Extension | Golimumab 200 mg Extension | Placebo - 50 mg Extension | Placebo - Golimumab100 mg Extension | Golimumab 50 mg - 100 mg Extension | Golimumab 100 mg - 200 mg Extension
Serious Adverse Events (participants affected / at risk) | 12/156 | 13/154 | 22/154 | 8/76 | 6/25 | 1/14 | 7/129 | 34/230 | 63/405 | 7/56 | 8/96 | 11/93 | 91/469 | 1/7 | 0/1 | 7/28 | 1/19 | 0/10
Other Adverse Events (participants affected / at risk) | 88/156 | 102/154 | 94/154 | 44/76 | 15/25 | 10/14 | 67/129 | 140/230 | 247/405 | 30/56 | 43/96 | 58/93 | 329/469 | 6/7 | 1/1 | 19/28 | 11/19 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance (N=156) | GLM-I-Rsp-Golimumab 50 mg Maintenance (N=154) | GLM-I-Rsp-Golimumab 100 mg Maintenance (N=154) | GLM-I-Rsp-Placebo Maintenance-Golimumab 100 mg (N=76) | GLM-I-Rsp-Golimumab 50 mg Maintenance-Golimumab 100 mg (N=25) | GLM-I-Rsp-Golimumab 100 mg Maintenance-Golimumab 200 mg (N=14) | Placebo Induction Responders (PBO-I-Rsp)-Placebo Maintenance (N=129) | PBO-I-nonRsp-Golimumab 100 mg Maintenance (N=230) | GLM-I-nonRsp-Golimumab 100 mg Maintenance (N=405) | PBO-I-Rsp-Placebo Maintenance-Golimumab 100 mg (N=56) | Placebo Extension (N=96) | Golimumab 50 mg Extension Phase (N=93) | Golimumab 100 mg Extension (N=469) | Golimumab 200 mg Extension (N=7) | Placebo - 50 mg Extension (N=1) | Placebo - Golimumab100 mg Extension (N=28) | Golimumab 50 mg - 100 mg Extension (N=19) | Golimumab 100 mg - 200 mg Extension (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia of Chronic Disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aplastic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Autoimmune Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Macular Fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 3 | 3 | 6 | 6 | 3 | 0 | 3 | 13 | 43 | 4 | 1 | 2 | 18 | 0 | 0 | 2 | 0 | 0
Colon Dysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Crohn's Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestinal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Volvulus of Small Bowel (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polyserositis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess Intestinal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disseminated Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Extrapulmonary Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Rotavirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Infected Cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infectious Colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Otitis Externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pilonidal Cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 6 | 0 | 0 | 0 | 0 | 0
Pneumonia Legionella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tick-Borne Viral Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Accidental Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penetrating Abdominal Trauma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spondylopathy Traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver Function Test Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seronegative Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Huerthle Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian Epithelial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Demyelination (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial Paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multiple Sclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nerve Root Compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Depression Suicidal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depressive Symptom (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Substance Abuse (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder Neck Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pelvi-Ureteric Obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine Polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal Prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity Vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lichen Sclerosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyoderma Gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic Aneurysm Rupture (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Golimumab Induction Responders (GLM-I-Rsp)-Placebo Maintenance (N=156) | GLM-I-Rsp-Golimumab 50 mg Maintenance (N=154) | GLM-I-Rsp-Golimumab 100 mg Maintenance (N=154) | GLM-I-Rsp-Placebo Maintenance-Golimumab 100 mg (N=76) | GLM-I-Rsp-Golimumab 50 mg Maintenance-Golimumab 100 mg (N=25) | GLM-I-Rsp-Golimumab 100 mg Maintenance-Golimumab 200 mg (N=14) | Placebo Induction Responders (PBO-I-Rsp)-Placebo Maintenance (N=129) | PBO-I-nonRsp-Golimumab 100 mg Maintenance (N=230) | GLM-I-nonRsp-Golimumab 100 mg Maintenance (N=405) | PBO-I-Rsp-Placebo Maintenance-Golimumab 100 mg (N=56) | Placebo Extension (N=96) | Golimumab 50 mg Extension Phase (N=93) | Golimumab 100 mg Extension (N=469) | Golimumab 200 mg Extension (N=7) | Placebo - 50 mg Extension (N=1) | Placebo - Golimumab100 mg Extension (N=28) | Golimumab 50 mg - 100 mg Extension (N=19) | Golimumab 100 mg - 200 mg Extension (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 5 | 2 | 1 | 0 | 2 | 10 | 22 | 1 | 2 | 1 | 20 | 1 | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 2 | 7 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 2 | 5 | 0 | 2 | 0 | 1 | 0 | 7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Eye Irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 10 | 11 | 3 | 2 | 0 | 5 | 9 | 21 | 0 | 4 | 6 | 28 | 0 | 1 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 4 | 1 | 1 | 0 | 1 | 2 | 2 | 6 | 0 | 1 | 3 | 11 | 0 | 1 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 29 | 25 | 18 | 7 | 2 | 1 | 17 | 25 | 49 | 7 | 20 | 17 | 111 | 2 | 0 | 7 | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 0 | 0 | 2 | 5 | 6 | 0 | 0 | 4 | 11 | 0 | 0 | 1 | 1 | 1
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 5 | 4 | 2 | 1 | 2 | 3 | 7 | 1 | 4 | 7 | 32 | 1 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 2 | 1 | 0 | 0 | 3 | 4 | 2 | 1 | 1 | 1 | 14 | 1 | 0 | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 1 | 5 | 0 | 0 | 0 | 5 | 1 | 4 | 0 | 2 | 3 | 10 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 3 | 3 | 1 | 1 | 1 | 3 | 4 | 7 | 0 | 2 | 3 | 13 | 0 | 0 | 1 | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 7 | 7 | 1 | 2 | 1 | 6 | 3 | 16 | 1 | 4 | 2 | 19 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 2 | 3 | 1 | 1 | 0 | 1 | 1 | 7 | 0 | 3 | 0 | 15 | 0 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 6 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 4 | 4 | 6 | 2 | 0 | 0 | 5 | 6 | 4 | 3 | 1 | 2 | 12 | 1 | 0 | 0 | 0 | 0
Feeling Cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 5 | 6 | 1 | 1 | 2 | 6 | 0 | 0 | 0 | 1 | 0
Injection Site Erythema (General disorders) | 1 | 1 | 4 | 3 | 0 | 1 | 1 | 3 | 5 | 0 | 0 | 1 | 7 | 1 | 0 | 2 | 0 | 0
Injection Site Induration (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection Site Rash (General disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 3 | 4 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 6 | 1 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 7 | 6 | 3 | 2 | 4 | 1 | 1 | 9 | 16 | 1 | 3 | 7 | 31 | 1 | 0 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Seasonal Allergy (Immune system disorders) | 3 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 1 | 0 | 3 | 11 | 1 | 0 | 1 | 1 | 0
Acute Tonsillitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 3 | 6 | 1 | 1 | 0 | 0 | 2 | 1 | 10 | 2 | 1 | 4 | 21 | 0 | 0 | 3 | 0 | 0
Chlamydial Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 4 | 1 | 0 | 0 | 3 | 5 | 0 | 0 | 0 | 0 | 0
Eyelid Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 2 | 3 | 2 | 0 | 0 | 2 | 4 | 4 | 1 | 0 | 5 | 23 | 0 | 0 | 2 | 0 | 2
Gastroenteritis Viral (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 3 | 4 | 0 | 0 | 2 | 8 | 2 | 0 | 1 | 0 | 0
Giardiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 1 | 14 | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 1 | 5 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 4 | 7 | 2 | 1 | 0 | 0 | 7 | 7 | 10 | 1 | 3 | 9 | 37 | 0 | 0 | 1 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 10 | 14 | 23 | 7 | 4 | 3 | 5 | 17 | 33 | 3 | 5 | 10 | 77 | 2 | 1 | 4 | 0 | 1
Oral Herpes (Infections and infestations) | 3 | 2 | 2 | 2 | 0 | 0 | 0 | 3 | 6 | 1 | 1 | 1 | 21 | 1 | 0 | 2 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 4 | 7 | 5 | 2 | 0 | 1 | 0 | 7 | 6 | 0 | 1 | 6 | 23 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 3 | 6 | 6 | 1 | 1 | 0 | 3 | 5 | 9 | 1 | 3 | 5 | 42 | 0 | 0 | 1 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Tinea Cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 4 | 1 | 0 | 0 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 8 | 8 | 6 | 3 | 1 | 6 | 16 | 20 | 4 | 4 | 6 | 39 | 1 | 0 | 2 | 2 | 2
Urinary Tract Infection (Infections and infestations) | 4 | 3 | 1 | 2 | 0 | 1 | 4 | 2 | 2 | 1 | 2 | 2 | 14 | 0 | 0 | 0 | 1 | 0
Viral Infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 3 | 4 | 2 | 2 | 3 | 9 | 1 | 0 | 1 | 1 | 0
Viral Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 4 | 4 | 0 | 1 | 1 | 11 | 2 | 0 | 0 | 0 | 0
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 4 | 0 | 0 | 1 | 0 | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0
Animal Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 1
Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 5 | 1 | 0 | 0 | 0 | 0
Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 3 | 3 | 0 | 0 | 0 | 3 | 6 | 6 | 0 | 0 | 2 | 7 | 0 | 0 | 1 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 5 | 2 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 1 | 6 | 0 | 0 | 1 | 0 | 1
Blood Calcium Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Blood Parathyroid Hormone Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 1 | 0 | 0 | 1 | 0
Neutrophil Count Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vitamin D Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White Blood Cell Count Increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 11 | 9 | 7 | 0 | 1 | 7 | 11 | 29 | 2 | 5 | 9 | 24 | 0 | 0 | 3 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7 | 1 | 0 | 1 | 5 | 6 | 10 | 1 | 1 | 2 | 30 | 0 | 0 | 2 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 1 | 0 | 1 | 0 | 5 | 2 | 0 | 0 | 1 | 7 | 0 | 0 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Demyelination (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 14 | 13 | 12 | 8 | 2 | 2 | 6 | 22 | 25 | 3 | 1 | 6 | 36 | 1 | 1 | 2 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 2 | 2 | 3 | 0 | 2 | 0 | 12 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 3 | 3 | 1 | 0 | 1 | 4 | 0 | 5 | 1 | 0 | 1 | 10 | 1 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 2 | 5 | 10 | 1 | 2 | 1 | 8 | 1 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Cervix Haemorrhage Uterine (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 8 | 1 | 0 | 0 | 5 | 10 | 18 | 2 | 8 | 4 | 36 | 0 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 0 | 1 | 9 | 0 | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 6 | 0 | 1 | 0 | 0 | 3 | 10 | 1 | 0 | 4 | 19 | 1 | 0 | 0 | 1 | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 4 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 4 | 0 | 0 | 2 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 3 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 7 | 1 | 0 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 9 | 6 | 1 | 0 | 1 | 2 | 7 | 11 | 2 | 1 | 3 | 16 | 1 | 0 | 0 | 1 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot Flush (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 4 | 1 | 1 | 0 | 0 | 0 | 1 | 5 | 11 | 2 | 0 | 3 | 12 | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
12 months after study ends, sponsor will be provided with a copy of the materials at least 45 days prior to submission, with details of proposed date, journal or conference name of publication & it will have 30 days post receipt to send a written request that the publication be delayed on the basis it exposes intellectual property that requires propriety protection but it will be only for 60 days after which investigator will be free to publish. The participation of sponsor will be acknowledged.